CLINICAL TRIAL: NCT06845098
Title: Impact of Thyroid Treatment on Ovarian Function and Pregnancy Outcomes in Women with Differentiated Thyroid Cancer: a Prospective Cohort Study
Brief Title: Impact of Thyroid Treatment on Ovarian Function and Pregnancy Outcomes in Women with Differentiated Thyroid Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024117-Ge
Record Dates: First submitted 2025-02-10; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Gland
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Thyroid one-sided lobe + isthmus resection (Experimental): Thyroid one-sided lobe + isthmus resection
  Interventions: Procedure: Thyroid one-sided lobe + isthmus resection
- Total thyroidectomy (Experimental): Total thyroidectomy
  Interventions: Procedure: Total thyroidectomy
- Total thyroidectomy + RAIT (Experimental): Total thyroidectomy + RAIT
  Interventions: Procedure: Total thyroidectomy + RAIT

INTERVENTIONS:
Procedure: Total thyroidectomy — Total thyroidectomy
  Arms: Total thyroidectomy
Procedure: Total thyroidectomy + RAIT — Total thyroidectomy + RAIT
  Arms: Total thyroidectomy + RAIT
Procedure: Thyroid one-sided lobe + isthmus resection — Thyroid one-sided lobe + isthmus resection
  Arms: Thyroid one-sided lobe + isthmus resection

SUMMARY:
This project aims to study the effects of different types of thyroid surgery and RAIT on ovarian function and pregnancy outcomes of DTC women of childbearing age, analyze possible risk factors, and assess whether potential risk factors such as age, thyroid stimulating hormone (TSH) levels and positive thyroid antibodies are related to ovarian hypofunction and adverse pregnancy outcomes.

DETAILED DESCRIPTION:
1) Screen the patients in the group according to the inclusion and exclusion criteria and sign the informed consent form (a total of 300 patients were included). Fill in the questionnaire after joining the group. 2) Physical examination of patients before treatment (measure height, weight, waist circumference, hip circumference, body fat distribution and percentage); thyroid function test (thyroid B-ultrasound, TSH, FT3, FT4, TPO-Ab, TG-Ab); baseline ovarian function test (AMH, menstruation 1-3 days Six hormones, observe the ovarian condition and the number of sinus follicles through vaginal B-ultrasound); leave blood for scientific research: 2 tubes of coagulation (serum), 1 tube of whole blood, -80℃ freeze. 3) Different types of thyroid surgery (thyroid unilateral lobe + isthmus resection, total thyroidectomy, total thyroidectomy + RAIT) are treated. 4) 3, 6, 12 and 24 months after treatment, the patients in the group should be followed up on ovarian and thyroid function, including physical examination (measurement of height, weight, waist circumference, hip circumference, body fat distribution and percentage); thyroid function testing (thyroid B-ultrasound, TSH, FT3, FT4, TPO-Ab, T G-Ab); ovarian function test (AMH, six items of sex hormones for 1-3 days of menstruation, observation of ovarian conditions and the number of sinus follicles through vaginal B-ultrasound); retention of blood for scientific research: 2 tubes (serum) of blood-promoting blood, 1 tube of whole blood, -80℃ freezing; record adverse reactions and combined medication. 5) If the patient in the group is pregnant during the follow-up period, the pregnancy follow-up shall be carried out according to the CRF table items at 2, 4, 12, 28 and 37 weeks of pregnancy respectively; delivery follow-up shall be carried out on the day of delivery and 6 weeks after delivery. 6) After the research, collect and sort out data for statistical analysis, summarize and sort out the results and publish them in professional journals in relevant fields in the form of papers.

ELIGIBILITY:
Inclusion criteria:

1. Age 20-45 years old;
2. Premenopausal women whose thyroid B-ultrasound + surgical pathology is clearly differentiated thyroid cancer (papillar thyroid cancer or follicular thyroid cancer);
3. TNM stage is in stage I (T1-3, N0 or N1, M0);
4. Treatment of thyroid tumor resection: unilateral lobe of the thyroid + isthmus resection, total thyroidectomy, total thyroidectomy + RAIT.

Exclusion criteria:

1. Patients with malignant tumors in other parts or low undifferentiated thyroid cancer;
2. Patients with abnormal liver and kidney function;
3. TNM stage II and above;
4. History of ovarian surgery, hysterectomy, pelvic surgery or radiation therapy;
5. Pregnancy;
6. Have the following uterine abnormalities, such as uterine malformation (single-horned uterus, double uterus); untreated mediastinal uterus, submucosal uterine fibroids, multiple endometrial polyps, or severe uterine adhesion.
7. Patients diagnosed with polycystic ovary syndrome by the Rotterdam standard;
8. Patients with ovarian failure;
9. Patients have infectious factors, immune diseases and metabolic diseases that may affect pregnancy outcomes;
10. Pregnancy contraindications or diseases that have a clear impact on pregnancy.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
AMH level | before treatment and 3, 6, 12 and 24 months after treatment
  Measure the concentration of AMH in serum

SECONDARY OUTCOMES:
Thyroid function | before tratment and 3, 6, 12 and 24 months after treatment
  Measure the level of TSH、T3、T4、FT3、FT4、TGAB、TPOAB in serum
clinical pregnancy rate | up to 24 months after the treatment
  Clinical pregnancy is defined as the detection of intrauterine gestational sac through ultrasound, and the clinical pregnancy rate is calculated by clinically pregnant women/total women.

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Ge, Study Chair — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No